CLINICAL TRIAL: NCT01696448
Title: Changes in Appetite, Weight, Body Composition, Endothelial Function and Biomarkers in Patients With the Cardiometabolic Syndrome: Comparison of a Combination of Berberine, Lipoic Acid, and Picrorhiza (CAR-191) Versus Placebo (The "BANGALORE" Study)
Brief Title: The BANGALORE Study; Combination of Berberine, Lipoic Acid, and Picrorhiza
Acronym: CAR-191
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carmel Biosciences (Industry)
Collaborators: Atlanta Vascular Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AVR-2012-01
Record Dates: First submitted 2012-08-13; First posted 2012-10-01 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Metabolic Syndrome
Keywords: Appetite Suppression; CAR-191
MeSH Terms: conditions — Metabolic Syndrome | interventions — Berberine; Thioctic Acid; Picrorhiza root extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (Experimental): CAR-191: Berberine 200mg, Alpha-lipoic Acid 150mg, Picrorhiza 100mg each in a separate capsule, to be taken 3 times a day, 30 minutes before breakfast, lunch and dinner. Total 9 capsules per day.
  Interventions: Dietary Supplement: CAR-191
- Control Group (Placebo Comparator): 3 placebo capsules, to be taken 3 times a day, 30 minutes before breakfast, lunch and dinner. Total 9 capsules per day.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: CAR-191 — Patients will be randomized to the CAR-191 intervention group in a 3:1, CAR0-191:placebo ratio. There will be 30 patients in the CAR-191 treatment group.
  Other Names: Berberine; Alpha-lipoic Acid; Picrorhiza
  Arms: Experimental Group
Other: Placebo — Patients will be randomised in a 3:1 ratio. There will be 10 patients in the placebo group.
  Arms: Control Group

SUMMARY:
Though medical treatment has been effective in the treatment of cardiometabolic diseases (including coronary atherosclerosis and diabetes mellitus), the incidence of these disorders continues to be high. Many reasons are responsible, but lifestyle changes, including an increased prevalence of obesity and the metabolic syndrome, are significant for this cause. Diagnosis and treatment of obese patients with hypertension requires that health care providers address the issues of hypertension, glucose intolerance, body weight and dyslipidemia. A sedentary lifestyle and poor cardiorespiratory fitness are not only associated with the (cardio) metabolic syndrome but could actually be considered features of the metabolic syndrome. These issues are significant in the health of certain individuals, who experience greater difficulty in treated BP control, experience increased hypertensive and diabetic complications, and have higher levels of obesity.

In this study, the investigators will evaluate the efficacy of the nutritional supplements berberine, alpha-lipoic acid, and picrorhiza (CAR-191) when consumed 30 minutes before meals, on appetite suppression, body composition and weight control. Additionally, the investigators will evaluate the effects of this combination of nutraceuticals on the mechanistic effects of oxidation, inflammation, and vascular function in a high-risk population with the metabolic syndrome.

Primary Objective To assess the comparative effect of a combination (known as CAR-191) of berberine (200 mg), alpha-lipoic acid (150 mg), and picrorhiza (100 mg) three times a day, compared to placebo three times a day, on parameters relate to appetite suppression, weight control and body composition in a high risk population with the metabolic syndrome.

Secondary Co-objectives

To evaluate the effects of CAR-191 versus placebo on changes in:

* Endothelial function using noninvasive brachial artery reactivity (BAR) ultrasound
* Biomarkers including IL-6, HOMA-IR, HbA1C, hsCRP, adiponectin, plasma/urine isoprostanes, PAI-1, TNFα-II, aldosterone, and glutathione redox ratio
* Urinary protein excretion
* Clinical chemistry including plasma glucose, blood urea nitrogen, creatinine, total bilirubin, uric acid, transaminases (SGOT/AST, SGPT/ALT), alkaline phosphatase, C-reactive protein, and lipoproteins

DETAILED DESCRIPTION:
Though medical treatment has been effective in the treatment of cardiometabolic diseases (including coronary atherosclerosis and diabetes mellitus), the incidence of these disorders continues to be high. Many reasons are responsible, but lifestyle changes, including an increased prevalence of obesity and the metabolic syndrome, are significant for this cause. Recent reported guidelines by the JNC-VII and National Cholesterol Education Panel/ATP-III suggest that blood pressure reduction is effective in improving the overall quality of life and may be helpful in the prevention of cardiovascular disease.

Diagnosis and treatment of obese patients with hypertension requires that health care providers address the issues of hypertension, glucose intolerance, body weight and dyslipidemia. Strategies to promote therapeutic lifestyle change (TLC), specifically increased physical activity and reduced dietary intake resulting in weight loss, are not as well defined. A sedentary lifestyle and poor cardiorespiratory fitness are not only associated with the (cardio) metabolic syndrome but could actually be considered features of the metabolic syndrome. These issues are significant in the health of certain individuals, who experience greater difficulty in treated BP control, experience increased hypertensive and diabetic complications, and have higher levels of obesity.

In this study, the investigators will evaluate the efficacy of the nutritional supplements berberine, alpha-lipoic acid, and picrorhiza (CAR-191) when consumed 30 minutes before meals, on appetite suppression, body composition and weight control. Additionally, the investigators will evaluate the effects of this combination of nutraceuticals on the mechanistic effects of oxidation, inflammation, and vascular function in a high-risk population with the metabolic syndrome.

The investigators will evaluate the initiation of CAR-191 in patients which meet at least 3 of the 5 criteria (ATP-III guidelines) for the cardiometabolic syndrome. The investigators will determine whether the CAR-191 combination as compared to placebo provides benefit in appetite suppression, body composition and certain clinical endpoints, including effects on endothelial function, lipid levels, and glucose control. This study will analyze the effects of 12 week administration of CAR-191 versus placebo on these parameters in a population of patients (n=40) with the cardiometabolic syndrome. The study has a parallel design consisting of 2 weeks of washout and then 12 weeks of treatment to either CAR-191 or placebo. The total study period is 14 weeks. Patients will be assigned to the CAR-191 or placebo group in a 3:1 ratio so that 30 patients will receive CAR-191 and 10 patients will receive placebo. See attached study design.

Primary Objective To assess the comparative effect of a combination (known as CAR-191) of berberine (200 mg), alpha-lipoic acid (150 mg), and picrorhiza (100 mg) three times a day, compared to placebo three times a day, on parameters relate to appetite suppression, weight control and body composition in a high risk population with the metabolic syndrome.

Secondary Co-objectives

To evaluate the effects of CAR-191 versus placebo on changes in:

* Endothelial function using noninvasive brachial artery reactivity (BAR) ultrasound
* Biomarkers including IL-6, HOMA-IR, HbA1C, hsCRP, adiponectin, plasma/urine isoprostanes, PAI-1, TNFα-II, aldosterone, and glutathione redox ratio
* Urinary protein excretion
* Clinical chemistry including plasma glucose, blood urea nitrogen, creatinine, total bilirubin, uric acid, transaminases (SGOT/AST, SGPT/ALT), alkaline phosphatase, C-reactive protein, and lipoproteins

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ≥ 18 years and ≤ 80 years with (cardio)metabolic syndrome as identified by investigators, OR
* Male and female subjects ≥ 18 years and ≤ 80 years with (cardio)metabolic syndrome defined by ATP-III criteria:

Insulin resistance, identified by 1 of the following

* Type 2 diabetes with HgA1C < 8.0% or on medical therapy
* Impaired fasting glucose
* Impaired glucose tolerance
* Or for those with normal fasting glucose levels (<100 mg/dl), glucose uptake below the lowest quartile for background population under investigation under hyperinsulinemic, euglycemic conditions

Plus any 2 of the following:

* Plasma triglycerides ≥ 150 mg/dl (≥ 1.7 mmol/L)
* HDL cholesterol <35 mg/dl (<0.9 mmol/L) in men or <39 mg/dl) (1.0 mmol/L) in women
* BMI >30 kg/m2 and/or waist:hip ratio > 0.9 in men, >0.85 in women
* Urinary albumin excretion rate ≥ 20 µg/min or albumin:creatinine ratio ≥ 30 mg/g

Exclusion Criteria:

* • Females of childbearing potential who are pregnant, lactating or who do not employ adequate birth control procedures.

  * Presence of any serious disorder including, renal, pulmonary, hepatic, gastrointestinal, endocrine/metabolic (with the exception of non-insulin dependent type 2 diabetes), hematologic/oncologic, neurologic and psychiatric diseases are exclusionary.
  * History of heart failure.
  * Stroke or heart attack within past 6 months.
  * Use of insulin.
  * Non-dominant upper arm circumference greater than 50 cm. (19.5 inches)
  * Currently using any prescription or over-the-counter weight loss products
  * Previous bariatric surgery or other weight reduction procedures
  * Weight loss or gain of greater than 15 pounds in the last 3 months
  * Past or current diagnosis of an eating disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-08; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
appetite suppression | 12 weeks
  Change in appetite will be measured through food frequency and appetite questionnaires

SECONDARY OUTCOMES:
Endothelial function using noninvasive brachial artery reactivity (BAR) ultrasound | 12 weeks
Weight control | 12 weeks
  Weight will be measured as body weight in lbs and BMI to see if treatment results in weight loss
Body Composition | 12 weeks
  Body composition will be measured as body fat percentage, fat mass, fat-free mass and waist to hip ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Syed T Rahman, MD, Principal Investigator — Atlanta Vascular Research Foundation
Locations (1):
- Atlanta Vascular Research Foundation, Atlanta, Georgia, United States